CLINICAL TRIAL: NCT02557347
Title: The Efficacy of Managing Fluid Overload in Peritoneal Dialysis Patient by a Structured Nurse-lead Intervention Protocol
Brief Title: Fluid Overload in Peritoneal Dialysis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Cheuk-Chun SZETO, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FO_in_PD
Record Dates: First submitted 2015-09-21; First posted 2015-09-23 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Aggressive fluid management
  Interventions: Behavioral: Aggressive fluid management

INTERVENTIONS:
Behavioral: Aggressive fluid management — nursing education, dietary advice, extra hypertonic dialysis cycles

SUMMARY:
The objective of this study is to determine the effectiveness of treating peritoneal dialysis (PD) patients with fluid overload by a structured nurse-lead intervention protocol. We plan to recruit 100 PD patients with fluid overload. These patients will be assessed and managed by a renal nurse specialist in the ambulatory renal center according to a standardized protocol. The improvement in the degree of overhydration will be determined by bioimpedance spectroscopy 4 and 12 weeks after treatment.

DETAILED DESCRIPTION:
Fluid overload is a common problem in peritoneal dialysis (PD) patients and it is associated with left ventricular hypertrophy and other adverse cardiac consequences. Fluid management is therefore an important aspect in the management of dialysis patient. In Hong Kong, PD patients with common medical problems related to dialysis are assessed and managed in the renal nurse clinic by pre-approved intervention protocols. Although it is the general impression that management of PD patients with fluid overload by a nurse-lead intervention protocol is robust and could reduce the work load of medical staff, the efficacy of this approach remains undetermined. The objective of this study is to determine the effectiveness of treating PD patients with fluid overload by a structured nurse-lead intervention protocol. We plan to recruit 100 PD patients with fluid overload, which is defined as overhydration (OH) ≥ 2 litres as measured by bioimpedance spectroscopy. These patients will be assessed and managed by a renal nurse specialist in the ambulatory renal center according to a standardized protocol previously approved by the Hospital Authority. The improvement in the degree of overhydration will be determined by bioimpedance spectroscopy 4 and 12 weeks after treatment. Change in body weight, blood pressure, degree of oedema, as well as the knowledge on salt and fluid restriction will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* PD patients with overhydration (OH) ≥ 2 litres as measured by bioimpedance spectroscopy

Exclusion Criteria:

* overt pulmonary edema and required urgent medical care
* cognitive impairment or problem of communication
* unlikely to survive for more than three months
* mechanical problems of the dialysis catheter
* active peritonitis or peritoneal failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
degree of overhydration | 12 weeks
  measured by bioimpedance spectroscopy

SECONDARY OUTCOMES:
blood pressure | 12 weeks
patient knowledge | 12 weeks
  questionnaire assessment

CONTACTS AND LOCATIONS:
Overall Officials: Cheuk Chun Szeto, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Renal Unit, Prince of Wales Hospital, Shatin, Hong Kong